CLINICAL TRIAL: NCT06181838
Title: Single-Blinded Randomized Controlled Trial: Comparison of Quality of Life in Moderate Acne Vulgaris Patients Based on Acne-QoL-INA Using Standard Therapy With and Without Acne Lesions Extraction
Brief Title: Comparison of Quality of Life in Moderate Acne Vulgaris Patients Based on Acne-QoL-INA Using Standard Therapy With and Without Acne Lesions Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Christa Desire Gracia, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 23-05-0571
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Acne Vulgaris; Quality of Life
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Standard therapy and lesion extraction
  Interventions: Procedure: Lesion extraction
- Control (Placebo Comparator): Standard therapy without lesion extraction
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Procedure: Lesion extraction — Tretinoin and benzoil peroxide used concurent in both groups as standard therapy
  Other Names: Tretinoin; Benzoil peroxide
  Arms: Intervention
Drug: Tretinoin — Tretinoin and benzoil peroxide used concurent in both groups as standard therapy
  Other Names: Benzoil peroxide
  Arms: Control

SUMMARY:
This study will compare the quality of life between 2 groups, which are group that receive standard moderate acne therapy in addition of lesion extractions, and the second group which only receive standard moderate acne therapy without lesion extractions.

DETAILED DESCRIPTION:
The group allocation will be randomized. Outcome of the study is the quality of life score based on Acne-QoL-INA questionnaire. The study duration is 8 weeks, consists of baseline visit and 2 follow ups at 4th and 8th weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as moderate acne vulgaris
* Able to read and speak in Indonesia
* Indonesian Citizen
* Sign the consent form

Exclusion Criteria:

* Pregnant of breastfeeding women
* Acne vulgaris lesion located only outside of face
* Experiencing COVID-19 symptoms
* Using retinoid acid containing cream or benzoil peroxide in the last 2 weeks
* Consume any oral antibiotics in the last 1 month
* Injected with intralesional steroid or having acne lesions extracted in the last 2 weeks
* Having laser or chemical peeling in the last 1 month

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Score | Every 4 weeks, measured until 8 weeks
  Measured using Acne-QoL-INA questionnaire

SECONDARY OUTCOMES:
Acne Grading | Every 4 weeks, measured until 8 weeks
  Lehmann classification of Acne Grading

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Umum Pusat Nasional Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia